CLINICAL TRIAL: NCT03336580
Title: A Phase 1, Open-label, Dose Escalation Study of Intravenous PRX004 in Subjects With Amyloid Transthyretin (ATTR) Amyloidosis
Brief Title: A Study of PRX004 in Subjects With Amyloid Transthyretin (ATTR) Amyloidosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Because of the impact of COVID-19 pandemic
Sponsor: Prothena Biosciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRX004-101; 2017-003521-15 (EudraCT Number)
Record Dates: First submitted 2017-10-23; First posted 2017-11-08 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Amyloidogenic Transthyretin (ATTR) Amyloidosis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Intervention Model Description: Dose Escalation Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRX004 (Experimental): Dose escalation in up to 6 dose levels
  Expansion of previously studied cohort(s) from Dose Escalation
  Extended dosing at RP2D
  Interventions: Drug: PRX004

INTERVENTIONS:
Drug: PRX004 — PRX004 (0.1, 0.3, 1, 3, 10, and 30 mg/kg) IV every 28 days
  PRX004 IV every 28 days at RP2D(s)
  PRX004 IV every 28 days at RP2D(s)

SUMMARY:
A Phase 1, open-label study of intravenous (IV) PRX004 as a single agent in subjects with hereditary amyloid transthyretin (hATTR) amyloidosis. The study will consist of 3 phases and will enroll up to a total of 36 subjects. A 3+3 dose escalation component to determine the safety, tolerability, PK, PD, and MTD. An expansion component in anticipated PRX004 RP2D cohorts selected from the Dose Escalation Phase. An extended dosing component for eligible subjects from the Dose Escalation or Expansion phases.

DETAILED DESCRIPTION:
This Phase 1, open-label consists of 3 phases. The Dose Escalation Phase is a 3+3 dose escalation component to determine the safety, tolerability, PK, PD, and MTD of IV PRX004 when given as a single agent in up to 36 evaluable subjects with hATTR amyloidosis. The Expansion Phase is an expansion component in anticipated PRX004 RP2D cohorts selected from the Dose Escalation Phase (this may occur in addition to cohorts in which additional subjects were added due to the observation of a dose-limiting [DLT] in the Escalation Phase). The Long-term Extension (LTE) Phase is an extended dosing component for eligible subjects from the Dose Escalation or Expansion phases.

The Dose Escalation Phase will follow a standard 3+3 design, in which cohorts of 3 to 6 subjects with hATTR amyloidosis will be enrolled at each dose level to receive IV PRX004 once every 28 days, based on scheduling from Month 1-Day 1 for up to 3 doses. Each subject will participate in only 1 dose escalation cohort. The starting dose of PRX004 will be 0.1 mg/kg.

Dose escalation will occur after the third evaluable subject in a cohort has completed the first 28 days following the first administration of PRX004. Up to 6 dose levels of PRX004 may be investigated (0.1, 0.3, 1, 3, 10, and 30 mg/kg) if tolerable. In the event the starting dose of 0.1 mg/kg is not tolerated, the dose escalationwill be halted and the study stopped.

Each subject will receive a maximum of 3 infusions of PRX004 in the Dose Escalation Phase. Subjects who complete the Month 3-Day 22 Visit in the Dose Escalation or Expansion phases may be eligible to receive up to 15 additional PRX004 infusions in the LTE Phase.

Each subject will receive a maximum of 3 infusions of PRX004 in the Dose Escalation Phase. Subjects who complete the Month 3-Day 22 Visit in the Dose Escalation or Expansion phases may be eligible to receive up to 15 additional PRX004 infusions in the LTE Phase.

Subjects who completed the EOS Visit in the Dose Escalation Phase prior to implementation of Protocol Amendment 2 may re-enter the study in the LTE Phase if they meet specific inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Ability to understand and willingness to sign an informed consent form prior to initiation of any study procedures
3. Diagnosis of amyloidosis determined by polarizing light microscopy of green birefringent material in Congo Red-stained tissue specimens; and confirmed diagnosis of ATTR amyloidosis by immunohistochemistry, mass spectrometry, documentation of an ATTR mutation by gene sequencing, or 99m technetium-3,3-diphosphono-1,2-propanodicarboxylic acid (99mTc-DPD) scans and/or technetium pyrophosphate (PYP) SPECT cardiac imaging. If scintigraphy is used for diagnosis then the grade must be 2 or greater, indicative of transthyretin amyloidosis-cardiomyopathy (ATTR-CM) (Gillmore, 2016)
4. Known TTR mutation
5. [Inclusion Criterion 5 removed in Amendment 2]
6. Patients receiving concomitant tafamidis or diflunisal may enroll in the study, providing the dose has been stable for the last 6 months
7. Karnofsky Performance Status (KPS) ≥60%
8. Adequate organ function, including all of the following:

   1. Adequate bone marrow reserve, defined as the following: absolute neutrophil count ≥1.0 × 109/L; platelet count ≥100 × 109/L; hemoglobin ≥10 g/dL
   2. Hepatic: total bilirubin ≤ 2 times the upper limit of normal (× ULN), transaminases (aspartate aminotransferase and/or alanine aminotransferase) ≤3 × ULN; alkaline phosphatase ≤5 × ULN
   3. Renal: estimated glomerular filtration rate (eGFR) ≥45 mL/min/1.73 m2
9. If currently receiving a diuretic, must have been on a stable dose for at least 4 weeks prior to the first dose of study drug
10. Systolic blood pressure ≥90 mmHg and ≤180 mmHg
11. Subjects with cardiomyopathy must have an NT-proBNP ≥650 pg/mL and ≤5000 pg/mL (ie, ≥76.9 pmol/L and ≤591 pmol/L) or evidence of septal wall thickening >1.2 cm on echocardiogram
12. Must have a biopsy unless data are available from a previous one. The biopsy may be taken from any tissue or organ affected by ATTR amyloidosis (eg, skin, lip, abdominal fat pad, salivary gland), at the Investigator's discretion. Nerve biopsies are not required.
13. Women of childbearing potential must have 2 negative pregnancy tests during Screening, the second within 24 hours prior to the first administration of study drug, and must agree to use highly effective physician-approved contraception from Screening to 90 days following the last study drug administration
14. Male subjects must be surgically sterile or must agree to use highly effective physician-approved contraception from Screening to 90 days following the last study drug administration
15. Polyneuropathy Disability (PND) Score ≤IIIB
16. Neuropathy Impairment Score (NIS) ≥5 and ≤130

Exclusion Criteria:

1. Amyloid light chain or other non-ATTR amyloidosis
2. Any past history of or present abuse of alcohol, diabetes, B12 or folate deficiencies, autoimmune diseases, hereditary disorders other than transthyretin (eg, Charcot-Marie-Tooth), uncontrolled hypothyroidism, or other etiologies for the peripheral neuropathy
3. Received prior liver transplant
4. Planned liver transplant during the study
5. Modified body mass index (mBMI) ≤600 kg/m2 × g/L
6. New York Heart Association (NYHA) Functional Class III-IV (Appendix 2)
7. LVEF ≤45%
8. Uncontrolled symptomatic orthostatic hypotension
9. Myocardial infarction, unstable or uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia, within 6 months prior to the first dose of study drug
10. Any history of clinically significant sinus pauses on ECG
11. Sinus pauses >3 seconds in the day or sinus pauses >5 seconds at night during the 48-hour pre-dose cardiac monitoring (ie, prior to first dose of study drug)
12. Arrhythmia requiring treatment diagnosed during the 48-hour pre-dose cardiac monitoring (ie, prior to first dose of study drug). Note: subject could be reconsidered for entry into the study if appropriate treatment is obtained
13. Hospitalized for heart failure within the 12 weeks prior to the first dose of study drug
14. Uncontrolled infection, or active malignancy with the exception of the following:

    * Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer
    * Low risk prostate cancer with Gleason score <7 and prostate specific antigen <10 mg/mL
    * Any other cancer from which the subject has been disease-free for ≥2 years
15. Clinically significant pleural effusion per Investigator (e.g., presence of pleural effusion ≥30% in either hemithorax)
16. History of Grade ≥3 hypersensitivity-associated AEs or hypersensitivities to other monoclonal antibodies or the excipients found in the PRX004 formulation
17. Known HIV infection or known hepatitis B or C virus carrier
18. Women who are pregnant or breastfeeding
19. Treatment with an investigational agent within 30 days or 5 half-lives (whichever is longer) prior to Month 1-Day 1
20. Any condition which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the Medical Monitor or Investigator unacceptably increase the subject's risk by participating in the study
21. Treatment with patisiran or inotersen within 90 days or 5 halflives (whichever is longer) prior to Month 1-Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of PRX004 | 28 days
  Maximum Tolerated Dose of PRX004
Number of subjects with treatment-emergent adverse events and clinically significant changes in ECGs, echocardiograms, cardiac telemetry, vital signs, and laboratory evaluations | 3 months
  Number of subjects with treatment-emergent adverse events and clinically significant changes in ECGs, echocardiograms, cardiac telemetry, vital signs, and laboratory evaluations

SECONDARY OUTCOMES:
PRX004 pharmacokinetic parameters - Cmin | 3 months
  Minimum observed concentration (Cmin) of PRX004 in plasma
PRX004 pharmacokinetic parameters -Cmax | 3 months
  Maximum observed concentration (Cmax) of PRX004 in plasma
PRX004 pharmacokinetic parameters - T1/2 | 3 months
  Terminal elimination half-life (T1/2) of PRX004 in plasma
PRX004 pharmacokinetic parameters -AUClast | 3 months
  Area under the concentration-time curve from time zero to the last quantifiable concentration time-point (AUClast) of PRX004 in plasma
PRX004 pharmacokinetic parameters -AUCtau | 3 months
  Area under the concentration-time curve over the dosing interval (AUCtau) of PRX004 in plasma
Immunogenicity indicators | 3 months
  Immunogenicity indicators: Anti-drug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Oregon Health and Science University, Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
- Centro Hospitalar do Porto, Porto, Portugal
- Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid, Spain
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capustin M, Frishman WH. Transthyretin Cardiac Amyloidosis and Novel Therapies to Treat This Not-so-rare Cause of Cardiomyopathy. Cardiol Rev. 2021 Sep-Oct 01;29(5):263-273. doi: 10.1097/CRD.0000000000000387. PMID 34397539